CLINICAL TRIAL: NCT02171286
Title: The Oncopanel Pilot (TOP) Study
Status: Completed | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: H14-01212
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer Metastatic; Advanced Non-Small Cell Lung Carcinoma; Advanced Melanoma; Gastrointestinal Stromal Tumors; Patients With Diagnosed Malignancies Being Considered for Clinical Trials
Keywords: KRAS; EGFR; BRAF; NRAS and HRAS; PIK3CA; RAS-RAF-MEK-MAPK; HER2; IDH1 and IDH2; ALK; TP53; c-KIT; STAT1&3; PDGFRA; Metastatic colorectal cancer; Advanced non-small cell lung cancer; Advanced melanoma; Gastrointestingal Struma Tumor; Candidate genes implicated as potential prognostic and predictive biomarkers in patients with solid tumours; Circulating Tumor DNA
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Hereditary Sensory and Autonomic Neuropathies; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood, plasma and tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment

SUMMARY:
The BCCA Oncopanel is a clinical assay being developed to determine genotype status of a prospectively defined set of genes.

The purpose of this pilot study is to assess the feasibility and effect on clinical-decision-making of the Oncopanel test. Eligible patients are those with advanced lung, colorectal, melanoma and GIST cancers and patients with diagnosed malignancies being considered for clinical trials.

DETAILED DESCRIPTION:
Somatic mutations in solid tumors represent an established means of characterizing malignancies for prognostic, diagnostic and therapeutic purposes. Mutations in EGFR, KRAS, BRAF, and KIT and PDGFRA genes direct therapy in patients with advanced lung, colorectal, melanoma, and GIST tumors, respectively. Known or novel mutations in other genes may also be of clinical significance but are not identified by current genotyping offered to BC Cancer Agency (BCCA) patients. Furthermore, numerous candidate genes have been implicated as potential prognostic and predictive biomarkers in patients with solid tumours. As such, the Oncopanel is a clinical assay being developed to determine genotype status of a prospectively defined set of genes. The following clinically relevant set of genes and exons are included in the Oncpanel: KRAS, EGFR, BRAF, NRAS and HRAS, PIK3CA Signal Transduction Pathway Genes, RAS-RAF-MEK-MAPK Pathway, HER2, IDH1 and IDH2, ALK, TP53, c-KIT, STAT1&3 and PDGFRA. Additional testing on the tumour material will also include analysis of specific gene variants associated with adverse events or response to therapy.

Numerous studies have documented the presence of circulating tumour DNA (ctDNA) among patients with advanced and early stage malignancies (20-22). The ability to diagnose standard cancer mutations with a blood-based assay (a "liquid biopsy") has not yet been established but presents obvious advantages. The emergence of "resistance" mutations arising in the metastatic tumor or throughout the course of therapy is well documented (21, 22). A blood biopsy may represent more accurate determination of the tumor's genetic features than archival DNA specimen. Adequate tissue specimens can be difficult to obtain from some patients with diagnosed malignancies, particularly lung cancer. A blood biopsy may represent a less invasive and timelier means of diagnosing both standard and translational cancer mutations.

ELIGIBILITY:
Patients with archival tumor tissue and a known history of invasive malignancies are eligible if they meet one or more of the following criteria:

* Advanced colorectal cancer and eligible for standard KRAS testing,
* Advanced non-small cell lung cancer and eligible for standard EGFR testing,
* Advanced melanoma and eligible for standard BRAF testing,
* Gastrointestinal stromal tumors (GISTs) eligible for standard c-KIT and PDGFRA testing,
* Being considered for potential eligibility in clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced colorectal cancer, non-small cell lung cancer and melanoma and candidates for clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of days between receipt of archival tumour tissue and generation of the OncoPanel Report | 10 business days

SECONDARY OUTCOMES:
Percent of cases in which a Oncopanel report is generated on a tumour specimen that has been received | 1 year

OTHER OUTCOMES:
Percent of cases in which a genotypic finding identified by the Oncopanel is repeated on standard clinical assay for the purpose of guiding subsequent therapy | 1 year
Percent of patients enrolled on an approved clinical trial related to Oncopanel results | 1 year
Concordance between Oncopanel results and ctDNA sequencing | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, MD, Principal Investigator — British Columbia Cancer Agency
Locations (5):
- Canada (5):
  - Abbotsford Centre, BC Cancer Agency, Abbotsford, British Columbia
  - BC Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Centre, BC Cancer Agency, Surrey, British Columbia
  - Vancouver Centre, BC Cancer Agency, Vancouver, British Columbia
  - Vancouver Island Centre, BC Cancer Agency, Victoria, British Columbia

REFERENCES:
- [Background] Dienstmann R, Dong F, Borger D, Dias-Santagata D, Ellisen LW, Le LP, Iafrate AJ. Standardized decision support in next generation sequencing reports of somatic cancer variants. Mol Oncol. 2014 Jul;8(5):859-73. doi: 10.1016/j.molonc.2014.03.021. Epub 2014 Apr 4. PMID 24768039
- [Background] Johnson DB, Dahlman KH, Knol J, Gilbert J, Puzanov I, Means-Powell J, Balko JM, Lovly CM, Murphy BA, Goff LW, Abramson VG, Crispens MA, Mayer IA, Berlin JD, Horn L, Keedy VL, Reddy NM, Arteaga CL, Sosman JA, Pao W. Enabling a genetically informed approach to cancer medicine: a retrospective evaluation of the impact of comprehensive tumor profiling using a targeted next-generation sequencing panel. Oncologist. 2014 Jun;19(6):616-22. doi: 10.1634/theoncologist.2014-0011. Epub 2014 May 5. PMID 24797823
- [Background] Gray SW, Hicks-Courant K, Cronin A, Rollins BJ, Weeks JC. Physicians' attitudes about multiplex tumor genomic testing. J Clin Oncol. 2014 May 1;32(13):1317-23. doi: 10.1200/JCO.2013.52.4298. Epub 2014 Mar 24. PMID 24663044
- [Background] Jimeno A, Messersmith WA, Hirsch FR, Franklin WA, Eckhardt SG. KRAS mutations and sensitivity to epidermal growth factor receptor inhibitors in colorectal cancer: practical application of patient selection. J Clin Oncol. 2009 Mar 1;27(7):1130-6. doi: 10.1200/JCO.2008.19.8168. Epub 2009 Jan 5. PMID 19124802
- [Background] Douillard JY, Oliner KS, Siena S, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Williams R, Rong A, Wiezorek J, Sidhu R, Patterson SD. Panitumumab-FOLFOX4 treatment and RAS mutations in colorectal cancer. N Engl J Med. 2013 Sep 12;369(11):1023-34. doi: 10.1056/NEJMoa1305275. PMID 24024839
- [Background] Shi Y, Au JS, Thongprasert S, Srinivasan S, Tsai CM, Khoa MT, Heeroma K, Itoh Y, Cornelio G, Yang PC. A prospective, molecular epidemiology study of EGFR mutations in Asian patients with advanced non-small-cell lung cancer of adenocarcinoma histology (PIONEER). J Thorac Oncol. 2014 Feb;9(2):154-62. doi: 10.1097/JTO.0000000000000033. PMID 24419411
- [Background] Lee CK, Brown C, Gralla RJ, Hirsh V, Thongprasert S, Tsai CM, Tan EH, Ho JC, Chu da T, Zaatar A, Osorio Sanchez JA, Vu VV, Au JS, Inoue A, Lee SM, Gebski V, Yang JC. Impact of EGFR inhibitor in non-small cell lung cancer on progression-free and overall survival: a meta-analysis. J Natl Cancer Inst. 2013 May 1;105(9):595-605. doi: 10.1093/jnci/djt072. Epub 2013 Apr 17. PMID 23594426
- [Background] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808
- [Background] Cancer Genome Atlas Research Network. Comprehensive genomic characterization of squamous cell lung cancers. Nature. 2012 Sep 27;489(7417):519-25. doi: 10.1038/nature11404. Epub 2012 Sep 9. PMID 22960745
- [Background] Ogino S, Lochhead P, Giovannucci E, Meyerhardt JA, Fuchs CS, Chan AT. Discovery of colorectal cancer PIK3CA mutation as potential predictive biomarker: power and promise of molecular pathological epidemiology. Oncogene. 2014 Jun 5;33(23):2949-55. doi: 10.1038/onc.2013.244. Epub 2013 Jun 24. PMID 23792451
- [Background] Marks JL, Gong Y, Chitale D, Golas B, McLellan MD, Kasai Y, Ding L, Mardis ER, Wilson RK, Solit D, Levine R, Michel K, Thomas RK, Rusch VW, Ladanyi M, Pao W. Novel MEK1 mutation identified by mutational analysis of epidermal growth factor receptor signaling pathway genes in lung adenocarcinoma. Cancer Res. 2008 Jul 15;68(14):5524-8. doi: 10.1158/0008-5472.CAN-08-0099. PMID 18632602
- [Background] Gandhi L, Bahleda R, Tolaney SM, Kwak EL, Cleary JM, Pandya SS, Hollebecque A, Abbas R, Ananthakrishnan R, Berkenblit A, Krygowski M, Liang Y, Turnbull KW, Shapiro GI, Soria JC. Phase I study of neratinib in combination with temsirolimus in patients with human epidermal growth factor receptor 2-dependent and other solid tumors. J Clin Oncol. 2014 Jan 10;32(2):68-75. doi: 10.1200/JCO.2012.47.2787. Epub 2013 Dec 9. PMID 24323026
- [Background] Borger DR, Tanabe KK, Fan KC, Lopez HU, Fantin VR, Straley KS, Schenkein DP, Hezel AF, Ancukiewicz M, Liebman HM, Kwak EL, Clark JW, Ryan DP, Deshpande V, Dias-Santagata D, Ellisen LW, Zhu AX, Iafrate AJ. Frequent mutation of isocitrate dehydrogenase (IDH)1 and IDH2 in cholangiocarcinoma identified through broad-based tumor genotyping. Oncologist. 2012;17(1):72-9. doi: 10.1634/theoncologist.2011-0386. Epub 2011 Dec 16. PMID 22180306
- [Background] Turcan S, Rohle D, Goenka A, Walsh LA, Fang F, Yilmaz E, Campos C, Fabius AW, Lu C, Ward PS, Thompson CB, Kaufman A, Guryanova O, Levine R, Heguy A, Viale A, Morris LG, Huse JT, Mellinghoff IK, Chan TA. IDH1 mutation is sufficient to establish the glioma hypermethylator phenotype. Nature. 2012 Feb 15;483(7390):479-83. doi: 10.1038/nature10866. PMID 22343889
- [Background] Yi ES, Boland JM, Maleszewski JJ, Roden AC, Oliveira AM, Aubry MC, Erickson-Johnson MR, Caron BL, Li Y, Tang H, Stoddard S, Wampfler J, Kulig K, Yang P. Correlation of IHC and FISH for ALK gene rearrangement in non-small cell lung carcinoma: IHC score algorithm for FISH. J Thorac Oncol. 2011 Mar;6(3):459-65. doi: 10.1097/JTO.0b013e318209edb9. PMID 21278610
- [Background] Choi YL, Soda M, Yamashita Y, Ueno T, Takashima J, Nakajima T, Yatabe Y, Takeuchi K, Hamada T, Haruta H, Ishikawa Y, Kimura H, Mitsudomi T, Tanio Y, Mano H; ALK Lung Cancer Study Group. EML4-ALK mutations in lung cancer that confer resistance to ALK inhibitors. N Engl J Med. 2010 Oct 28;363(18):1734-9. doi: 10.1056/NEJMoa1007478. PMID 20979473
- [Background] Doebele RC, Pilling AB, Aisner DL, Kutateladze TG, Le AT, Weickhardt AJ, Kondo KL, Linderman DJ, Heasley LE, Franklin WA, Varella-Garcia M, Camidge DR. Mechanisms of resistance to crizotinib in patients with ALK gene rearranged non-small cell lung cancer. Clin Cancer Res. 2012 Mar 1;18(5):1472-82. doi: 10.1158/1078-0432.CCR-11-2906. Epub 2012 Jan 10. PMID 22235099
- [Background] Lux ML, Rubin BP, Biase TL, Chen CJ, Maclure T, Demetri G, Xiao S, Singer S, Fletcher CD, Fletcher JA. KIT extracellular and kinase domain mutations in gastrointestinal stromal tumors. Am J Pathol. 2000 Mar;156(3):791-5. doi: 10.1016/S0002-9440(10)64946-2. PMID 10702394
- [Background] Guo J, Si L, Kong Y, Flaherty KT, Xu X, Zhu Y, Corless CL, Li L, Li H, Sheng X, Cui C, Chi Z, Li S, Han M, Mao L, Lin X, Du N, Zhang X, Li J, Wang B, Qin S. Phase II, open-label, single-arm trial of imatinib mesylate in patients with metastatic melanoma harboring c-Kit mutation or amplification. J Clin Oncol. 2011 Jul 20;29(21):2904-9. doi: 10.1200/JCO.2010.33.9275. Epub 2011 Jun 20. PMID 21690468
- [Background] Carvajal RD, Antonescu CR, Wolchok JD, Chapman PB, Roman RA, Teitcher J, Panageas KS, Busam KJ, Chmielowski B, Lutzky J, Pavlick AC, Fusco A, Cane L, Takebe N, Vemula S, Bouvier N, Bastian BC, Schwartz GK. KIT as a therapeutic target in metastatic melanoma. JAMA. 2011 Jun 8;305(22):2327-34. doi: 10.1001/jama.2011.746. PMID 21642685
- [Background] Lu HF, Yang JS, Lin YT, Tan TW, Ip SW, Li YC, Tsou MF, Chung JG. Diallyl disulfide induced signal transducer and activator of transcription 1 expression in human colon cancer colo 205 cells using differential display RT-PCR. Cancer Genomics Proteomics. 2007 Mar-Apr;4(2):93-7. PMID 17804871
- [Background] Corless CL, Schroeder A, Griffith D, Town A, McGreevey L, Harrell P, Shiraga S, Bainbridge T, Morich J, Heinrich MC. PDGFRA mutations in gastrointestinal stromal tumors: frequency, spectrum and in vitro sensitivity to imatinib. J Clin Oncol. 2005 Aug 10;23(23):5357-64. doi: 10.1200/JCO.2005.14.068. Epub 2005 May 31. PMID 15928335
- [Background] Punnoose EA, Atwal S, Liu W, Raja R, Fine BM, Hughes BG, Hicks RJ, Hampton GM, Amler LC, Pirzkall A, Lackner MR. Evaluation of circulating tumor cells and circulating tumor DNA in non-small cell lung cancer: association with clinical endpoints in a phase II clinical trial of pertuzumab and erlotinib. Clin Cancer Res. 2012 Apr 15;18(8):2391-401. doi: 10.1158/1078-0432.CCR-11-3148. Epub 2012 Apr 5. PMID 22492982
- [Background] Spindler KL, Pallisgaard N, Vogelius I, Jakobsen A. Quantitative cell-free DNA, KRAS, and BRAF mutations in plasma from patients with metastatic colorectal cancer during treatment with cetuximab and irinotecan. Clin Cancer Res. 2012 Feb 15;18(4):1177-85. doi: 10.1158/1078-0432.CCR-11-0564. Epub 2012 Jan 6. PMID 22228631
- [Background] Misale S, Yaeger R, Hobor S, Scala E, Janakiraman M, Liska D, Valtorta E, Schiavo R, Buscarino M, Siravegna G, Bencardino K, Cercek A, Chen CT, Veronese S, Zanon C, Sartore-Bianchi A, Gambacorta M, Gallicchio M, Vakiani E, Boscaro V, Medico E, Weiser M, Siena S, Di Nicolantonio F, Solit D, Bardelli A. Emergence of KRAS mutations and acquired resistance to anti-EGFR therapy in colorectal cancer. Nature. 2012 Jun 28;486(7404):532-6. doi: 10.1038/nature11156. PMID 22722830
- [Background] Thompson JD, Shibahara G, Rajan S, Pel J, Marziali A. Winnowing DNA for rare sequences: highly specific sequence and methylation based enrichment. PLoS One. 2012;7(2):e31597. doi: 10.1371/journal.pone.0031597. Epub 2012 Feb 15. PMID 22355378
- [Background] Pel J, Broemeling D, Mai L, Poon HL, Tropini G, Warren RL, Holt RA, Marziali A. Nonlinear electrophoretic response yields a unique parameter for separation of biomolecules. Proc Natl Acad Sci U S A. 2009 Sep 1;106(35):14796-801. doi: 10.1073/pnas.0907402106. Epub 2009 Aug 17. PMID 19706437
- [Background] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- [Background] Green RC, Berg JS, Grody WW, Kalia SS, Korf BR, Martin CL, McGuire AL, Nussbaum RL, O'Daniel JM, Ormond KE, Rehm HL, Watson MS, Williams MS, Biesecker LG; American College of Medical Genetics and Genomics. ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. Genet Med. 2013 Jul;15(7):565-74. doi: 10.1038/gim.2013.73. Epub 2013 Jun 20. PMID 23788249